CLINICAL TRIAL: NCT00433875
Title: A Double-Blind, Placebo Controlled, Randomized, Parallel-Group Clinical Trial With Multiple Dose Treatment of Anti-IL 15 Human Monoclonal Antibody (AMG 714) in Patients With Active Rheumatoid Arthritis Who Have Previously Failed One or More Disease Modifying Anti-Rheumatic Drugs
Brief Title: Phase 2 AMG 714 in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030210
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — AMG-714

INTERVENTIONS:
Drug: AMG 714

SUMMARY:
Twelve week treatment of AMG 714 in RA patients who failed at least one DMARD, followed by a 3 month observational period.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of RA -

Exclusion Criteria: No prior biologic treatment for RA

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com